CLINICAL TRIAL: NCT06486857
Title: Accuracy Validation Study of a Novel Gas Detection Method for Dyslipidemia
Brief Title: Accuracy Assessment of a Novel Gas Detection Approach in Dyslipidemia Diagnosis
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KS2024055
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Dyslipidemias; Gas Detection Method
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — exhaled breath condensate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: a novel gas detection method for dyslipidemia screening — Multidimensional Mass Spectrometry Technologies Based on Exhaled Metabolic Fingerprint Spectra for Dyslipidemia Detection

SUMMARY:
This study aims to validate the feasibility and accuracy of a novel gas detection method for dyslipidemia screening by analyzing the lipid profile of human breath metabolites. It explores a simple, rapid, and non-invasive method for screening dyslipidemia. The application prospects of this method are broad; it can be used not only for early screening and monitoring of dyslipidemia in hospitals and communities, providing strong support for the prevention of cardiovascular diseases, but also for the routine monitoring and treatment effectiveness evaluation of patients with hyperlipidemia, offering a scientific basis for personalized treatment plans. This study not only has profound scientific value but also provides a theoretical basis for the development of subsequent new clinical testing methods.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Voluntarily signed the informed consent form

Exclusion Criteria:

1. Patients with lung cancer, asthma, chronic obstructive pulmonary disease, pulmonary cystic fibrosis, or acute respiratory distress syndrome
2. Women who are pregnant or breastfeeding
3. Patients with chronic kidney disease (GFR < 60 ml/min) or cirrhosis
4. Individuals unable to cooperate with the collection of exhaled gas samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
accuracy of cholesterol testing | within 1 week day of sample collection

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No